CLINICAL TRIAL: NCT06299488
Title: Combined Effects of Prunus Cerasus (Montmorency Tart Cherry) and Apocynum Venetum (Venetron®) On Sleep and Anxiety in Adults With Insomnia
Brief Title: Combined Effects of Prunus Cerasus and Apocynum Venetum On Sleep and Anxiety in Adults With Insomnia
Acronym: Sip2Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakshmi Nutraceuticals LLC (Industry)
Collaborators: People Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PS03
Record Dates: First submitted 2024-02-28; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Insomnia
Keywords: Sleep; Herbal; Sleep Aid
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Participants will complete a 5-week study consisting of screening assessments, baseline scales and surveys, objective digital measure, 2 weeks of product use (1 week on - 1 week off - 1 week on), scales and surveys, and end of study assessments and surveys. This is a remote observational study that will use the People Science app-based data collection platform Consumer Health Learning and Organizing Ecosystem (CHLOE) for study participants to report their assessments and collect objective sleep data from personal wearable devices. Participants will receive the study product during the baseline period. Demographic and medical history data will be collected for the study.
Masking Description: This study is not blinded. Participants consume the intervention on alternating weeks. All participants receive the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Montmorency Cherry + Apocynum Venetum (Experimental): Sip2Sleep® is a proprietary formula of Montmorency tart cherry extract and Venetron®, a purified, powdered extract derived from Apocynum Venetum. Recommended dose is ¼ teaspoon which contains 553 mg (1:5 fruit extract) of Montmorency tart cherry and 25mg of Venetron® leaf extract. The compound was prepared as an oral dropper, consumed alone or in water 30-60 minutes prior to bedtime. The study was conducted over a period of four weeks, consisting of two weeks without intervention and two weeks with intervention as follows: (1 week off (baseline) - 1 week on - 1 week off - 1 week on) for each participant
  Interventions: Other: Sip2Sleep: Montmorency Cherry and Apocynum Venetum
- No intervention: Typical Sleep Routine (No Intervention): The study was conducted over a period of four weeks, consisting of two weeks without intervention and two weeks with intervention (ABAB) as follows: (1 week off (baseline) - 1 week on - 1 week off - 1 week on) for each participant.
  Participants did not consume any intervention or placebo during this time.

INTERVENTIONS:
Other: Sip2Sleep: Montmorency Cherry and Apocynum Venetum — See arm description
  Arms: Intervention: Montmorency Cherry + Apocynum Venetum

SUMMARY:
Lay Summary: This study is about the effect of using a unique formula called Sip2Sleep®, a product currently available on the market which is a combination of montmorency tart cherry extract and Venetron® (Apocynum venetum leaf extract) on sleep. The purpose of this study is to evaluate the effects of taking this combination product on various aspects of sleep. This study is being conducted by People Science, and is sponsored by Lakshmi Nutraceuticals, LLC. The information we gather will help inform how people may use Sip2Sleep® to affect the quality of sleep.

Participants in this study will complete a number of surveys about their difficulties falling asleep and staying asleep (insomnia), their energy level during the day and health status regarding their quality of sleep.

There are no major risks associated with this study.

DETAILED DESCRIPTION:
The rationale for this study is to determine the effect of a consumer-grade, unique formula called Sip2Sleep®, which is a combination of Montmorency tart cherry extract and Venetron®, a patented, purified, powdered extract derived from the Rafuma leaf, Apocynum venetum, on sleep disturbance in adults. Because this product is currently available in the OTC market across the United States, a consumer-driven, decentralized observational clinical research study is well-suited for examining the effect of this formulation on sleep.

Sleep disturbance is highly prevalent and impacted by many interdependent variables. We will examine self-reported sleep disturbance in a broad age-range of adults who have chosen to use this product. The study will incorporate participant reported outcome questionnaires, daily surveys, and the participants' personal health tracking wearable device (e.g. Apple Watch, Fitbit, Smartwatch, etc.) to engage the participant in their sleep health and explore objective digital outcome measures of sleep. An important feature of this consumer-driven study design is to help individual consumers observe the effects of this product on their own sleep patterns during the study itself. There is no "doctor-patient" relationship as part of this research since the participant as a consumer is making the informed choice to take the product and take part in the observational process with self-reported measures. Findings from this study will contribute knowledge toward the design of future sleep research studies, the improvement of the Sip2Sleep® product formulation, and may help inform clinical recommendations for adults interested in using alternative products for sleep.

The following self-reporting measures are used in order to evaluate the effect of Sip2Sleep® in adults with self-reported sleep disturbance:

Surveys to reflect sleep quality, sleep latency, total sleep duration and level of alertness during the day to be distributed daily. Sleep quality and level of alertness during the day will be evaluated with a single 10-point visual analogue scale (VAS) and objective sleep data reflecting sleep latency and total sleep duration will be collected from personal wearable devices.

Insomnia Sleep Index (ISI) is a brief self-report instrument measuring the patient's perception of both nocturnal and diurnal symptoms of insomnia during the past two weeks. The ISI comprises seven items assessing the perceived severity of difficulties initiating sleep, staying asleep, and early morning awakenings, satisfaction with current sleep pattern, interference with daily functioning, noticeability of impairment attributed to the sleep problem, and degree of distress or concern caused by the sleep problem. Each item is rated on a five-point scale and the total score indicates the severity of insomnia, with a range of possible scores from 0-28. A score higher than 14 has been indicated to be the optimal cut-off for insomnia as a disorder. The ISI has been widely used in clinical and research settings as it is brief and easy to administer, and can provide valuable information for diagnosis and treatment planning. Research has found that the ISI is sensitive in detecting changes in the patient's perception of treatment outcome, and a good degree of convergence exists between the patient and the clinician's evaluation of insomnia severity.13,14 Generalized Anxiety Disorder-7 (GAD-7) is a self-reported anxiety survey utilized in primary care consisting of a 7-item anxiety scale. The instrument is well supported to use in a general population and normative data can be used to compare a subject's GAD-7 score with those determined from a general population reference group, with evidence of significant reliability and validity with congruent agreement in self-reported and interviewer-administered versions of the scale. GAD and Depression symptoms frequently occur together, but previous studies have supported via factor analysis that this measure can detect GAD and depression as distinct dimensions.15 This measure will be used in combination with other scales to observe self-reported effects on sleep disturbances and insomnia, such as anxiety or other psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Has self-reported sleep disturbance
* Insomnia Severity Index (ISI) score of > 15 at screening
* Interested in understanding more about the quality of their sleep and chose to use the Sip2Sleep product for sleep
* Willingness to do a minimum of 1 week wash out of current OTC or other products for sleep (e.g. melatonin, anticholinergics)
* Willingness to do a minimum of 1 week wash out of any cannabis products
* Able to receive shipment of the product at an address within the United States If taking prescription hypnotics (e.g. zolpidem, zaleplon, benzodiazepines) or other class of medication for sleep, must be on a stable dose for at least 4 weeks.
* Able to read and understand English
* Able to use a personal smartphone
* Has and is able to use a personal health tracking wearable device (e.g., Apple Watch, Fitbit Smartwatch, Oura Ring, etc.)
* Able to understand and provide informed consent
* Able to complete study assessments over 5 weeks

Exclusion Criteria:

* Research participants who have no computer, smartphone, and internet access and/or do not use a computer or smartphone
* The following concomitant therapies are excluded:
* Participants taking daily prescription medication for sleep (for example, prescription hypnotics like zolpidem, zaleplon, benzodiazepines) not on a stable dose for at least 4 weeks
* Participants receiving Cognitive Behavioral Therapy for Insomnia (CBTi)
* Participants receiving any investigational therapies or treatments
* Other Illnesses or Conditions: Participants who have the following co-morbidities are excluded:
* Confirmed diagnoses of the following sleep disorders: Narcolepsy, Restless Leg Syndrome, Circadian Rhythm Disorders
* Confirmed diagnosis of Sleep Apnea that is untreated or not well controlled
* Current or prior psychotic disorder
* Current or prior Substance Abuse Disorder
* Current or prior cardiac dysrhythmias (for example, atrial fibrillation, supraventricular tachycardia)
* Currently pregnant, planning to become pregnant in the next 1 month, or breastfeeding
* Allergies or adverse reactions (for example, anxiety) to Montmorency tart cherry extract and/or Venetron®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Subjective Sleep Quality | 14 days of no intervention versus 14 days of intervention use in a 28 day period, consisting of 1 Week on, 1 week off, 1 week on, 1 week off. Entire study completion for all participants within 1 year.
  Change in average sleep quality score by 1 point as measured by daily 10-point visual analogue rating scale (VAS) from baseline and 1 week of no product use

SECONDARY OUTCOMES:
Insomnia Sleep Index | 14 days of no intervention versus 14 days of intervention use in a 28 day period, consisting of 1 Week on, 1 week off, 1 week on, 1 week off. Entire study completion for all participants within 1 year.
  Change in Insomnia Sleep Index (ISI) by at least 4 points or more from baseline and 1 week of no product use
Generalized Anxiety Disorder-7 (GAD-7) | 14 days of no intervention versus 14 days of intervention use in a 28 day period, consisting of 1 Week on, 1 week off, 1 week on, 1 week off. Entire study completion for all participants within 1 year.
  Change in Generalized Anxiety Disorder-7 (GAD-7) by 4 points or more from baseline and 1 week of no product use
Subjective Alertness | 14 days of no intervention versus 14 days of intervention use in a 28 day period, consisting of 1 Week on, 1 week off, 1 week on, 1 week off. Entire study completion for all participants within 1 year.
  Change in average level of alertness during the daytime score by 1 point as measured by daily 10-point visual analogue rating scale (VAS)

OTHER OUTCOMES:
Exploratory: Sleep Duration | 14 days of no intervention versus 14 days of intervention use in a 28 day period, consisting of 1 Week on, 1 week off, 1 week on, 1 week off. Entire study completion for all participants within 1 year.
  Change in average nightly sleep duration as measured via personal health tracking wearable device
Exploratory: Sleep Latency | 14 days of no intervention versus 14 days of intervention use in a 28 day period, consisting of 1 Week on, 1 week off, 1 week on, 1 week off. Entire study completion for all participants within 1 year.
  Change in average nightly sleep latency as measured via personal health tracking wearable device
Participant Satisfaction | End of study survey, after completing the 28 study days
  Assessment of patient satisfaction survey of study experience including design and use of app-based data collection tools

CONTACTS AND LOCATIONS:
Overall Officials: Noah Craft, MD/PhD, Principal Investigator — People Science, Inc.
Locations (1):
- People Science Inc., West Hollywood, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foley L. Sleep Foundation: Insomnia.
- [Background] Losso JN, Finley JW, Karki N, Liu AG, Prudente A, Tipton R, Yu Y, Greenway FL. Pilot Study of the Tart Cherry Juice for the Treatment of Insomnia and Investigation of Mechanisms. Am J Ther. 2018 Mar/Apr;25(2):e194-e201. doi: 10.1097/MJT.0000000000000584. PMID 28901958
- [Background] Pigeon WR, Carr M, Gorman C, Perlis ML. Effects of a tart cherry juice beverage on the sleep of older adults with insomnia: a pilot study. J Med Food. 2010 Jun;13(3):579-83. doi: 10.1089/jmf.2009.0096. PMID 20438325
- [Background] Grundmann O, Nakajima J, Seo S, Butterweck V. Anti-anxiety effects of Apocynum venetum L. in the elevated plus maze test. J Ethnopharmacol. 2007 Apr 4;110(3):406-11. doi: 10.1016/j.jep.2006.09.035. Epub 2006 Oct 13. PMID 17101250
- [Background] Yang, J. et al. 2009. Safety study of Apocynum venetum extract in healthy adults. Journal of Nutritional Food, no. 12:1-9.
- [Background] Vissiennon C, Nieber K, Kelber O, Butterweck V. Route of administration determines the anxiolytic activity of the flavonols kaempferol, quercetin and myricetin--are they prodrugs? J Nutr Biochem. 2012 Jul;23(7):733-40. doi: 10.1016/j.jnutbio.2011.03.017. Epub 2011 Aug 12. PMID 21840194

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT06299488/Prot_SAP_000.pdf